CLINICAL TRIAL: NCT02610270
Title: Erythrocyte Omega-3 Fatty Acid Content in Elite Athletes in Response to Omega-3 Supplementation: A Dose-Response
Brief Title: Erythrocyte Omega-3 Fatty Acid Content in Elite Athletes
Acronym: O3Sport
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre d'Alt Rendiment (Other)
Responsible Party: Principal Investigator, FRANCISCO DROBNIC, MD, PhD, MD PhD, Centre d'Alt Rendiment
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CAR-2
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Sport; fatty acid; omega 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 Gums (Experimental): Athletes that continued their usual training and diet, who took 2 gums of omega 3 (DHA 760 mg) during the experimental period.
  Interventions: Dietary Supplement: 2 Gums
- 3 Gums (Experimental): Athletes that continued their usual training and diet, who took 3 gums of omega 3 (DHA 1140 mg) during the experimental period.
  Interventions: Dietary Supplement: 3 Gums
- Control (No Intervention): Athletes and coaches that continued their usual training and diet, but did not take any supplements during the experimental period.

INTERVENTIONS:
Dietary Supplement: 2 Gums — 760 mg DHA
  Arms: 2 Gums
Dietary Supplement: 3 Gums — 1140 mg DHA
  Arms: 3 Gums

SUMMARY:
A suitable concentration of omega-3 fatty acids in relation to omega 6 is considered necessary for a good cell function and prevention of various inflammatory processes. Diet and supplementation are the fundamental procedures to achieve the reference values for several years. Athletes are individuals under physical stress and higher tissue restoration, while maintaining adequate diets they show, as the rest of humans, lower than desired levels. In the present study the investigators aims to determine the modification of those levels by the administration of two different doses of a given product, keeping the same model of diet and physical and competition.

DETAILED DESCRIPTION:
The study aims to assess concentrations of the different fatty acids in the erythrocyte membrane before and after administration of a compound with high quality omega3 (EPA and DHA) in two different doses, compared with control group . The period of evaluation and management is four months, one month for the proposed renewal of red blood cells. The composition of the diet, the sports calendar, caloric expenditure and level of training is determined. During the study process it is excluded subjects with injuries or disease processes and ensure that no one take any supplement or modify workouts or diet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young men and women athletes from the Olympic Training Center (OTC) of Sant Cugat del Valles in Barcelona (Spain) (20 to 45 years of age) belonging to different summer sport activities were asked to participate.

Exclusion Criteria:

* Any type of inflammatory process, or the use of anti-inflammatory medications, consumption of n-3 Fatty Acids (FA) supplements and n-3 FA-supplemented foods in the past 3 months; planning to change dietary habits, or training schedule.
* During the study, any subject that falls under injury or need nonsteroidal antiinflammatory drug or get sick by inflammatory or infectious disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
fatty acid levels at the membrane of the red blood cells | Four months
  Evaluation will be obtained before and after the experimental period

SECONDARY OUTCOMES:
Impregnation in relation to dosage administrated to the athletes | Four months
  Evaluate the impregnation level of the membrane of red blood cells, taken into account the two dosages in relation of the subjects characteristics, sex (M,F), omega3 index (EPA/DHA%), weight (kg), age(years), etc. looking for a relationships of better or worse impregnation depending on sex, body weight, body mass index, previous level of omega3, etc.
Different level of impregnation of the red blood cells in relation to dosage and weight of the athletes | Four months
  Evaluate the impregnation level of the membrane of red blood cells, taken into account the two dosages in relation of the subjects characteristics, weight (kg).
Different level of impregnation of the red blood cells in relation to dosage and different previous omega 3 index of the athletes | Four months
  Evaluate the impregnation level of the membrane of red blood cells, taken into account the two dosages in relation of the subjects characteristic of previous level of omega3 index (EPA/DHA%)
Different level of impregnation of the red blood cells in relation to dosage and different sex of the athletes | Four months
  Evaluate the impregnation level of the membrane of red blood cells, taken into account the two dosages in relation of the sex (M,F) of the subjects
Different level of impregnation of the red blood cells in relation to dosage and different age of the athletes | Four months
  Evaluate the impregnation level of the membrane of red blood cells, taken into account the two dosages in relation of the age(years) of the subjects etc.

CONTACTS AND LOCATIONS:
Overall Officials: Franchek Drobnic, MD PhD, Principal Investigator — Olympic Training Center, Centre d'Alt Rendiment CAR

REFERENCES:
- [Background] Luchtman DW, Song C. Cognitive enhancement by omega-3 fatty acids from child-hood to old age: findings from animal and clinical studies. Neuropharmacology. 2013 Jan;64:550-65. doi: 10.1016/j.neuropharm.2012.07.019. Epub 2012 Jul 27. PMID 22841917
- [Background] Michael-Titus AT, Priestley JV. Omega-3 fatty acids and traumatic neurological injury: from neuroprotection to neuroplasticity? Trends Neurosci. 2014 Jan;37(1):30-8. doi: 10.1016/j.tins.2013.10.005. Epub 2013 Nov 22. PMID 24268818
- [Background] Yates CM, Calder PC, Ed Rainger G. Pharmacology and therapeutics of omega-3 polyunsaturated fatty acids in chronic inflammatory disease. Pharmacol Ther. 2014 Mar;141(3):272-82. doi: 10.1016/j.pharmthera.2013.10.010. Epub 2013 Nov 4. PMID 24201219
- [Background] Mickleborough TD. Omega-3 polyunsaturated fatty acids in physical performance optimization. Int J Sport Nutr Exerc Metab. 2013 Feb;23(1):83-96. doi: 10.1123/ijsnem.23.1.83. PMID 23400626
- [Background] Bloomer RJ, Larson DE, Fisher-Wellman KH, Galpin AJ, Schilling BK. Effect of eicosapentaenoic and docosahexaenoic acid on resting and exercise-induced inflammatory and oxidative stress biomarkers: a randomized, placebo controlled, cross-over study. Lipids Health Dis. 2009 Aug 19;8:36. doi: 10.1186/1476-511X-8-36. PMID 19691834
- [Background] Lewis EJ, Radonic PW, Wolever TM, Wells GD. 21 days of mammalian omega-3 fatty acid supplementation improves aspects of neuromuscular function and performance in male athletes compared to olive oil placebo. J Int Soc Sports Nutr. 2015 Jun 18;12:28. doi: 10.1186/s12970-015-0089-4. eCollection 2015. PMID 26085822
- [Background] Bailes JE, Patel V. The potential for DHA to mitigate mild traumatic brain injury. Mil Med. 2014 Nov;179(11 Suppl):112-6. doi: 10.7205/MILMED-D-14-00139. PMID 25373094
- [Background] Hasadsri L, Wang BH, Lee JV, Erdman JW, Llano DA, Barbey AK, Wszalek T, Sharrock MF, Wang HJ. Omega-3 fatty acids as a putative treatment for traumatic brain injury. J Neurotrauma. 2013 Jun 1;30(11):897-906. doi: 10.1089/neu.2012.2672. Epub 2013 Jun 5. PMID 23363551
- [Background] Di Girolamo FG, Situlin R, Mazzucco S, Valentini R, Toigo G, Biolo G. Omega-3 fatty acids and protein metabolism: enhancement of anabolic interventions for sarcopenia. Curr Opin Clin Nutr Metab Care. 2014 Mar;17(2):145-50. doi: 10.1097/MCO.0000000000000032. PMID 24500439
- [Background] Skulas-Ray AC. Omega-3 fatty acids and inflammation: a perspective on the challenges of evaluating efficacy in clinical research. Prostaglandins Other Lipid Mediat. 2015 Jan-Mar;116-117:104-11. doi: 10.1016/j.prostaglandins.2015.02.001. Epub 2015 Feb 16. PMID 25698680
- [Background] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005
- [Background] Enns JE, Yeganeh A, Zarychanski R, Abou-Setta AM, Friesen C, Zahradka P, Taylor CG. The impact of omega-3 polyunsaturated fatty acid supplementation on the incidence of cardiovascular events and complications in peripheral arterial disease: a systematic review and meta-analysis. BMC Cardiovasc Disord. 2014 May 31;14:70. doi: 10.1186/1471-2261-14-70. PMID 24885361
- [Background] von Schacky C, Kemper M, Haslbauer R, Halle M. Low Omega-3 Index in 106 German elite winter endurance athletes: a pilot study. Int J Sport Nutr Exerc Metab. 2014 Oct;24(5):559-64. doi: 10.1123/ijsnem.2014-0041. Epub 2014 Sep 8. PMID 25203220
- [Background] Delodder F, Tappy L, Liaudet L, Schneiter P, Perrudet C, Berger MM. Incorporation and washout of n-3 PUFA after high dose intravenous and oral supplementation in healthy volunteers. Clin Nutr. 2015 Jun;34(3):400-8. doi: 10.1016/j.clnu.2014.07.005. Epub 2014 Jul 15. PMID 25066733
- [Background] Flock MR, Skulas-Ray AC, Harris WS, Etherton TD, Fleming JA, Kris-Etherton PM. Determinants of erythrocyte omega-3 fatty acid content in response to fish oil supplementation: a dose-response randomized controlled trial. J Am Heart Assoc. 2013 Nov 19;2(6):e000513. doi: 10.1161/JAHA.113.000513. PMID 24252845
- [Background] Walker CG, Browning LM, Mander AP, Madden J, West AL, Calder PC, Jebb SA. Age and sex differences in the incorporation of EPA and DHA into plasma fractions, cells and adipose tissue in humans. Br J Nutr. 2014 Feb;111(4):679-89. doi: 10.1017/S0007114513002985. Epub 2013 Sep 24. PMID 24063767
- [Background] Welch RW, Antoine JM, Berta JL, Bub A, de Vries J, Guarner F, Hasselwander O, Hendriks H, Jakel M, Koletzko BV, Patterson CC, Richelle M, Skarp M, Theis S, Vidry S, Woodside JV; International Life Sciences Institute Europe Functional Foods Task Force. Guidelines for the design, conduct and reporting of human intervention studies to evaluate the health benefits of foods. Br J Nutr. 2011 Nov;106 Suppl 2:S3-15. doi: 10.1017/S0007114511003606. PMID 22129662
- [Background] Katan MB, Deslypere JP, van Birgelen AP, Penders M, Zegwaard M. Kinetics of the incorporation of dietary fatty acids into serum cholesteryl esters, erythrocyte membranes, and adipose tissue: an 18-month controlled study. J Lipid Res. 1997 Oct;38(10):2012-22. PMID 9374124
- [Background] Harris WS, Mozaffarian D, Lefevre M, Toner CD, Colombo J, Cunnane SC, Holden JM, Klurfeld DM, Morris MC, Whelan J. Towards establishing dietary reference intakes for eicosapentaenoic and docosahexaenoic acids. J Nutr. 2009 Apr;139(4):804S-19S. doi: 10.3945/jn.108.101329. Epub 2009 Feb 25. PMID 19244379
- [Background] Aranceta J, Perez-Rodrigo C. Recommended dietary reference intakes, nutritional goals and dietary guidelines for fat and fatty acids: a systematic review. Br J Nutr. 2012 Jun;107 Suppl 2:S8-22. doi: 10.1017/S0007114512001444. PMID 22591906
- [Background] Gomez Candela C, Bermejo Lopez LM, Loria Kohen V. Importance of a balanced omega 6/omega 3 ratio for the maintenance of health: nutritional recommendations. Nutr Hosp. 2011 Mar-Apr;26(2):323-9. doi: 10.1590/S0212-16112011000200013. PMID 21666970
- [Background] Skulas-Ray AC, Kris-Etherton PM, Harris WS, Vanden Heuvel JP, Wagner PR, West SG. Dose-response effects of omega-3 fatty acids on triglycerides, inflammation, and endothelial function in healthy persons with moderate hypertriglyceridemia. Am J Clin Nutr. 2011 Feb;93(2):243-52. doi: 10.3945/ajcn.110.003871. Epub 2010 Dec 15. PMID 21159789
- [Background] Browning LM, Walker CG, Mander AP, West AL, Madden J, Gambell JM, Young S, Wang L, Jebb SA, Calder PC. Incorporation of eicosapentaenoic and docosahexaenoic acids into lipid pools when given as supplements providing doses equivalent to typical intakes of oily fish. Am J Clin Nutr. 2012 Oct;96(4):748-58. doi: 10.3945/ajcn.112.041343. Epub 2012 Aug 29. PMID 22932281
- [Background] Tartibian B, Maleki BH, Abbasi A. The effects of omega-3 supplementation on pulmonary function of young wrestlers during intensive training. J Sci Med Sport. 2010 Mar;13(2):281-6. doi: 10.1016/j.jsams.2008.12.634. Epub 2009 Jun 12. PMID 19523875
- [Background] Arterburn LM, Hall EB, Oken H. Distribution, interconversion, and dose response of n-3 fatty acids in humans. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1467S-1476S. doi: 10.1093/ajcn/83.6.1467S. PMID 16841856
- [Background] Drobnic F, CordobillaB, Rueda F, Domingo JC. Caracterización de diferentes suplementos de ácidos omega-3 en su aplicación en las edades pediátricas Acta Pediatr Esp. 2013; 71(11): e353-e357
- [Background] Cao J, Schwichtenberg KA, Hanson NQ, Tsai MY. Incorporation and clearance of omega-3 fatty acids in erythrocyte membranes and plasma phospholipids. Clin Chem. 2006 Dec;52(12):2265-72. doi: 10.1373/clinchem.2006.072322. Epub 2006 Oct 19. PMID 17053155
- [Background] Flock MR, Harris WS, Kris-Etherton PM. Long-chain omega-3 fatty acids: time to establish a dietary reference intake. Nutr Rev. 2013 Oct;71(10):692-707. doi: 10.1111/nure.12071. Epub 2013 Oct 3. PMID 24117792
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Lemaitre RN, Tanaka T, Tang W, Manichaikul A, Foy M, Kabagambe EK, Nettleton JA, King IB, Weng LC, Bhattacharya S, Bandinelli S, Bis JC, Rich SS, Jacobs DR Jr, Cherubini A, McKnight B, Liang S, Gu X, Rice K, Laurie CC, Lumley T, Browning BL, Psaty BM, Chen YD, Friedlander Y, Djousse L, Wu JH, Siscovick DS, Uitterlinden AG, Arnett DK, Ferrucci L, Fornage M, Tsai MY, Mozaffarian D, Steffen LM. Genetic loci associated with plasma phospholipid n-3 fatty acids: a meta-analysis of genome-wide association studies from the CHARGE Consortium. PLoS Genet. 2011 Jul;7(7):e1002193. doi: 10.1371/journal.pgen.1002193. Epub 2011 Jul 28. PMID 21829377
- [Derived] Drobnic F, Rueda F, Pons V, Banquells M, Cordobilla B, Domingo JC. Erythrocyte Omega-3 Fatty Acid Content in Elite Athletes in Response to Omega-3 Supplementation: A Dose-Response Pilot Study. J Lipids. 2017;2017:1472719. doi: 10.1155/2017/1472719. Epub 2017 Jun 1. PMID 28656110